CLINICAL TRIAL: NCT05213533
Title: Kanagawa Intravenous and Endovascular Treatment Registry for Acute Ischemic Stroke
Brief Title: Kanagawa Intravenous and Endvascular Treatment Registry
Acronym: K-NET
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: St. Marianna University Toyoko Hospital (Other)
Responsible Party: Principal Investigator, Toshihiro Ueda, MD, Professor, Department of Strokology; Director, Stroke Center, St. Marianna University Toyoko Hospital
Other Study IDs: 3757
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Acute Ischemic Stroke
Keywords: acute stroke, mechanical thrombectomy, intravenous tPA
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The K-NET registry is a prospective, multicenter, observational registry study for all consecutive patients who received intravenous tPA therapy and/or endovascular treatment for acute ischemic stroke. This study is attended by 40 of the 58 Primary Stroke Centers in Kanagawa Prefecture, which is located in the Tokyo metropolitan area and has a population of 9.24 million. Patient enrollment for this study began in January 2018.

DETAILED DESCRIPTION:
Inclusion criteria for this study are all consecutive patients who meet either or both of the patients who received intravenous tPA therapy for acute ischemic stroke and intention to perform EVT for large vessel occlusion. There were no exclusion criteria. The local neurologists, neurosurgeons, and neurointerventionalists at each institution made the decision to perform EVT and intravenous tPA.

The primary outcome was good as defined by the modified Rankin Scale (mRS) of 0 to 2 at three months. We also determined a favorable outcome: mRS 0-2 or not worsening of the mRS score at three months. Secondary analyses included predicting a favorable outcome using multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for this study are all consecutive patients who meet either or both of the patients who received intravenous tPA therapy for acute ischemic stroke and intention to perform EVT for large vessel occlusion.

Exclusion Criteria:

There were no exclusion criteria. There are no upper or lower age limits for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Kanagawa prefecture in Japan
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | after 3 months
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 6. This is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months following hospital discharge.
  0 The patient has no residual symptoms.
  1. The patient has no significant disability; able to carry out all pre-stroke activities.
  2. The patient has slight disability; unable to carry out all pre-stroke activities but able to look after self without daily help.
  3. The patient has moderate disability; requiring some external help but able to walk without the assistance of another individual.
  4. The patient has moderately severe disability; unable to walk or attend to bodily functions without assistance of another individual.
  5. The patient has severe disability; bedridden, incontinent, requires continuous care.
  6. The patient has expired.

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiro Ueda, MD, Principal Investigator — St. Marianna University Toyoko Hospital
Locations (1):
- St.Marianna University Toyoko Hospital, Kawasaki, Kanagawa, Japan

REFERENCES:
- [Derived] Ueda T, Hasegawa Y, Takeuchi M, Morimoto M, Yamamoto R, Tsuboi Y, Kaga Y, Ito H, Onodera H, Takaishi S, Tatsuno K, Usuki N, Yoshie T, Murata H, Yamano Y; K-NET Registry Investigators. Comparative analysis of outcome-associated factors following endovascular treatment for intracranial atherosclerotic disease and cardioembolism: A subanalysis of the K-NET registry. Interv Neuroradiol. 2025 Aug 1:15910199251361304. doi: 10.1177/15910199251361304. Online ahead of print. PMID 40746094